CLINICAL TRIAL: NCT05097924
Title: Gastrointestinal Tolerability of a Partially Hydrolyzed, Whey-based, Ready-to-feed Infant Formula in Healthy Newborns During the Birth Hospitalization Period: a Post-market Study
Brief Title: Gastrointestinal Tolerability of a Partially Hydrolyzed Ready-to-feed Infant Formula in Healthy Newborns
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 21.07.INF
Record Dates: First submitted 2021-10-04; First posted 2021-10-28 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Infant Nutritional Physiological Phenomena; Infant Formula

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: NAN Supreme HypoAllergenic Starter Infant Formula in ready-to-feed format — Post-market observational study with formula feeding administered via standard of care

SUMMARY:
Gastrointestinal tolerability of a partially hydrolyzed, whey-based, ready-to-feed infant formula in healthy newborns during the birth hospitalization period: a post-market study

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained from both parents or a legally acceptable representative (LAR).
* Full-term gestational birth (≥ 37 completed weeks of gestation), with a birth weight of ≥ 2500 g and ≤ 4500 g.
* Parent(s) must have independently elected, before enrollment, to formula feed.
* Infant age ≤ 24 hours after birth.
* Child's parents / LAR are of legal age of consent, must understand the informed consent form and other study documents, and are willing and able to fulfill the requirements of the study protocol.

Exclusion Criteria:

* Infant is exclusively breastfed.
* Evidence of significant cardiac, respiratory, endocrine, hematologic, gastrointestinal, or other systemic diseases, infections, or disorders.
* Infant has other condition that, in the judgement of the investigator, would make the infant inappropriate for entry into the study.
* Conditions that require infant feedings other than those specified in the protocol.
* Infant is currently participating in another interventional clinical trial that impacts study outcomes.

Ages: 0 Months to 24 Months | Sex: All
Age Groups: Child
Study Population: Newborn infants
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Parent-reported individual gastrointestinal (GI) symptoms and GI-related behaviors | Daily through study completion (age 2 to 5 days)
  The Newborn Infant GI Tolerance eDiary will be completed daily (preferably in the evening) by parents, who will document the frequency and severity of diarrhea, gassiness, spitting-up, vomiting, reflux, abdominal pain, fussiness, crying, and sleep patterns using a 6-point scale (from Never to Always). Higher scores indicate more symptoms of GI discomfort.
Parent-reported individual GI- and feeding-related behaviors | At study completion (age 2 to 5 days)
  At discharge, parents will complete the Gastrointestinal Tract Function sub-scale of the NeoEAT questionnaire (either the Bottle-Feeding or the Mixed-Feeding version, depending on the mother's chosen feeding mode) to document GI- and feeding-related behaviors using a 6-point scale (from Never to Always). Higher scores indicate more symptoms of GI discomfort and problematic feeding behavior.
Number of infants with specific GI characteristics | Daily through study completion (age 2 to 5 days)
  GI symptoms and GI-related behaviors, as documented by health care providers in the infants' hospital medical charts (e.g., diarrhea, constipation, and vomiting)
Number of feeds per day | Daily through study completion (age 2 to 5 days)
  Number of formula feeds per day, number of breastfeeds per day (if mixed fed), as documented by health care providers in the infants' hospital medical charts

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Sulaiman Al Habib Hospital, Riyadh, Saudi Arabia